CLINICAL TRIAL: NCT00758381
Title: A Randomized Phase II Study of Gemcitabine/Cisplatin With or Without Sorafenib to Evaluate the Efficacy and Safety in Patients With Locally Advanced or Metastatic Pancreatic Cancer. MAPS Trial
Brief Title: Metastatic Advanced Pancreas Sorafenib
Acronym: MAPS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gruppo Italiano per lo studio dei Carcinomi dell'Apparato Digerente (Other)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Stefano CASCINU, Medical Professor, Fondazione GISCAD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-001781-32
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2008-10-10 (Estimated); Status verified 2008-10

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: pancreatic cancer; advanced or metastatic; sorafenib
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm Metastasis | interventions — Sorafenib; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Sorafenib 400 mg po bid, continuously
  Gemcitabine 1000 mg/m2, Cisplatin 25 mg/m2 day 1, and 8 every 21 days.
  Interventions: Drug: Sorafenib 400 mg po bid, continuously
- B (Active Comparator): Gemcitabine 1000 mg/m2, Cisplatin 25 mg/m2 day 1, and 8 every 21 days
  Interventions: Drug: Gemcitabina, Cisplatino

INTERVENTIONS:
Drug: Sorafenib 400 mg po bid, continuously — NEXAVAR*112CPR RIV 200MG
  Titolare AIC:
  BAYER SpA
  Numero di AIC dell'IMP:
  037154010
  Other Names: L01XE05 V; Sostanza attiva o descrizione del livello ATC selezionato; SORAFENIB TOSILATO
  Arms: A
Drug: Gemcitabina, Cisplatino — Gemcitabina 1000 mg/mq, Cisplatino 25 mg/mq day 1 and 8 every 21 days
  Other Names: GEMZAR*INFUS 1FL 1G POLV; Titolare AIC:; ELI LILLY ITALIA SpA; Numero di AIC dell'IMP:; 029452012; CISPLATINO TEVA*EV 50MG 100ML; TEVA PHARMA ITALIA Srl; 026543025
  Arms: B

SUMMARY:
This is multicentre, open-label, randomized, phase II trial in patients with locally advanced or metastatic pancreatic cancer. Subjects will be randomized in a 1:1 ratio to receive gemcitabine/cisplatin in combination with Sorafenib (arm A) or gemcitabine/cisplatin alone (arm B), as first-line chemotherapy.

DETAILED DESCRIPTION:
Up to date no standard treatment is available for pancreatic cancer. Although gemcitabine is commonly used in patients with pancreatic cancer with the purpose of symptom palliation, there is no clear evidence of efficacy in terms of survival increase or progression control. Furthermore, attempts at improving results by combining gemcitabine with other cytotoxic drugs failed to obtain any advantage. Recently, an EGFR inhibitor (erlotinib) showed a small survival advantage when combined with gemcitabine. results obtained with a combination of gemcitabine and oxaliplatin seem more promising. A meta-analysis of randomised trials comparing gemcitabine versus gemcitabine and platinum analogues showed a statistical significant survival advantage for the combination.

Sorafenib is an inhibitor of the RAS/RAF signalling pathway. Furthermore, sorafenib is able to inhibit both VEGFR and PDGFR.

Since RAS and RAF mutations are quite common in pancreatic cancer, Sorafenib could be useful in the management of these tumours. Furthermore, it may be combined with gemcitabine and cisplatin without any pharmacokinetic interaction or enhanced toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to beginning protocol specific procedures
* Male or female 18 to 75 years of age
* Diagnosis of histologically confirmed adenocarcinoma of the pancreas
* Locally advanced (non-resectable) or metastatic pancreatic cancer
* Presence of at least one uni-dimensional indicator lesion measurable by CT scan or MRI in not an irradiated area (RECIST criteria)
* Karnofsky performance status of ≥ 70 at study entry
* Neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L, and hemoglobin ≥ 9 g/dL
* Bilirubin level either normal or < 1.5 x ULN
* ASAT and ALAT ≤ 2.5 X ULN (≤ 5 x ULN if liver metastasis are present)
* Serum creatinine < 1.5 x ULN
* Amylase and lipase ≤ 1.5 x the upper limit of normal
* PT or INR and PTT < 1.5 x upper limit of normal (subjects who receive anti-coagulation treatment with an agent such as warfarin or heparin will be allowed to participate provided that no evidence of underlying abnormality in these parameters exists).
* Effective contraception for both male and female patients if the risk of conception exists

Exclusion Criteria:

* Brain metastases
* Previous chemotherapy for locally advanced or metastatic pancreatic cancer.
* Adjuvant therapy if documented recurrence is within 6 months after the end of adjuvant treatment)
* Radiotherapy within 4 weeks prior to study entry
* Major surgery within 4 weeks of first dose of study drug
* Concurrent chronic systemic immune therapy
* Any investigational agent(s) 4 weeks prior to entry
* Clinically relevant coronary artery disease or a history of a myocardial infarction within the last 6 months
* Thrombotic or embolic events such as cerebrovascular accident including transient ischemic attacks within the past 6 months
* Acute or subacute intestinal occlusion or history of inflammatory bowel disease
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited legal capacity
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent
* Women who are pregnant or breastfeeding
* Acute or subacute intestinal occlusion
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 5 years will be allowed to enter the trial).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | time from randomization date to date of local or regional relapse

SECONDARY OUTCOMES:
- overall Response Rate (RECIST Criteria) - duration of response - overall survival time | time from the day of randomization to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Cascinu, M.Professor, Study Chair — GISCAD Foundation
Locations (17):
- Italy (17):
  - A.O. Universitaria Ospedali Riuniti Umberto I, Ancona, Ancona
  - Ospedali Riuniti, Largo Barozzi, 1, Bergamo, Bergamo
  - A.O. Treviglio-Caravaggio, P.le Ospedale n1, Treviglio, Bergamo
  - A.O.Policlinico S.Orsola Malpighi, Bologna, Bologna
  - Ospedale S.Orsola Fatebenefratelli, Brescia, BS
  - A.O. Careggi-Università, Viale Pieraccini, 17, Florence, Firenze
  - Ospedale Galliera, Genova, Genova
  - A.O. Ospedale S.Martino, Genova, GE
  - A.O. Carlo Poma - Via Albertoni, 1, Mantova, Mantova
  - A.O. Cà Granda, Piazza Ospedale Maggiore, 3, Milan, Milano
  - A.O. san Paolo, Milan, MI
  - Casa di Cura Igea, Milan, MI
  - Ospedale S.Carlo Borromeo, Milan, MI
  - A.O. S.Gerardo, Monza, MI
  - Policlinico di modena, Modena, Modena
  - Università Campus Biomedico, Via Emilio Longoni, 83, Roma, Roma
  - A.O. S.Giovanni Calabita Fatebenefratelli, Roma, Roma